CLINICAL TRIAL: NCT00646204
Title: A 16 Week, Investigator-initiated, Single-center, Double Blind, Randomized, Placebo-controlled Trial of Namenda® (Memantine Hcl) for Non-motor Symptoms in Parkinson's Disease
Brief Title: Namenda (Memantine) for Non-motor Symptoms in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Joseph Jankovic, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-18912
Record Dates: First submitted 2007-12-28; First posted 2008-03-28 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; non-motor symptoms
MeSH Terms: conditions — Parkinson Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Active study drug (Experimental): memantine 10 mg bid
  Interventions: Drug: Memantine
- 2-placebo comparator (Placebo Comparator): 2 tabs bid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Memantine — 10 mg bid
  Other Names: Namenda
  Arms: 1-Active study drug
Drug: placebo — 2 tabs bid
  Arms: 2-placebo comparator

SUMMARY:
To evaluate the effects of Memantine on non-motor symptoms in patients with Parkinson's disease.

Parkinson's disease (PD) affects about one million people in the United States. It is a common neurological condition that is clinically defined by rigidity (muscle stiffness), bradykinesia (slowness of movement) and tremor. Parkinson's Disease , however, reveals numerous non-motor symptoms that have been underemphasized. Problematic symptoms include varying degrees of dementia, psychosis, diminished assertiveness and confidence, general fatigue, excessive daytime sleepiness, problems with blood pressure, sweating, and bladder, and a common yet difficult to define sense of "not feeling well".

DETAILED DESCRIPTION:
Patients were enrolled over 11 months from the Parkinson Disease Center and Movement Disorder Clinic at Baylor College of Medicine. PD was diagnosed using standard criteria. Specific inclusion criteria were intentionally broad and included both fluctuating and non-fluctuating patients with a UPDRS "motivation" (#4) score of greater or equal to 2. Patients with dementia (MMSE<24) or taking amantadine were excluded.

The patients signed an informed consent approved by the Baylor College of Medicine Institutional Review Board and the study was registered on Clinical Trials.gov #NCT00646204. The study was funded by a grant from the Forest Research Institute.

After baseline assessments, patients (N=40) were randomized equally to drug (N=20) and placebo (N=20) groups. This was done by a computerized random number generator by a coordinator not otherwise involved in the study.

Patients completed medical and medication histories, a Unified Parkinson's Disease Rating Scale (UPDRS), a battery of neuropsychiatric assessments (see Table 2), global impressions, and adverse events. Patients were not allowed to change other PD medications. The drug/placebo dosing began at 5 mg/day and increased to 5 mg 2x/day, 10 mg / 5 mg, and finally 10 mg 2x/day, in weekly increments. After a safety call (2 weeks after initiation) they returned for identical assessments at week 8. Drug accountability was documented at each visit. An 8-week open label extension was started if desired using the same protocol and assessments.

Tabulations and univariate statistics on difference scores between visits were run using Intercooled Stata V8.0 for windows (Stata Corporation, College Station, Texas 77845), and included Student's t-test with equal variances and contingency table analysis using Pearson's Chi-square test. Statistics were done using LOCF. Corrections for multiple comparisons were not done.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between the ages of 18 and 80 inclusive.
2. Each subject must meet standard criteria for PD.
3. All patients on dopaminergic therapy must report benefit. -No other abnormal neurological signs. -No direct or indirect trauma to the nervous system within 3 months preceding the onset of PD. -No convincing evidence of sudden onset or evidence of stepwise deterioration.
4. Subjects must be in generally good health as evidenced by previous medical history and clinical examination.
5. Subjects will be allowed to take any PD medication with the exception of amantadine. They will also be allowed to take medications approved for the use of Alzheimer's disease.
6. Subjects will be required to be on a stable dose of all medications for at least two weeks prior to entry into the study and may not alter these medications throughout the study.
7. If subjects are on an anti-depressant medications, a stable dose of these will be required for at least six weeks prior to entry into the study.
8. Subjects must be accessible by telephone.
9. If the subject is a female of childbearing age, she must have had: a hysterectomy, or tubal ligation, or otherwise be incapable or pregnancy, or have practiced one of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide and barrier, intrauterine device, partner sterility.
10. Female of childbearing age must have had a negative urine pregnancy test within one week of study entry. 11. Prior to participation in this study, each subject must sign an informed consent.

Exclusion Criteria:

1. Subjects who do not meet inclusion criteria.
2. Subjects who are not able to abstain from alcohol for 24 hours prior to each evaluation.
3. Subjects who can not maintain an identical dose of any medicine that may affect PD symptoms or signs during their entire study involvement.
4. Subjects who have exhibited meaningful psychiatric disease not thought to be related to PD. (Depression and psychosis typical for PD will not be excluded). 5. Subjects who have previously taken memantine.

6. Subjects currently taking Amantadine. 7. Subjects with greater than moderate dementia (MMSE<24). 8. Subjects with co-morbid disease that in the investigators decision could interfere with treatment with memantine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Ondo, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- PDCMDC 6550 Fannin, Suite 1801, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No individual data available

REFERENCES:
- [Background] Ondo WG, Shinawi L, Davidson A, Lai D. Memantine for non-motor features of Parkinson's disease: a double-blind placebo controlled exploratory pilot trial. Parkinsonism Relat Disord. 2011 Mar;17(3):156-9. doi: 10.1016/j.parkreldis.2010.12.003. Epub 2010 Dec 30. PMID 21193343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After baseline assessments, patients (N=40) were randomized to drug and placebo groups. They received a battery of neuropsychiatric assessments. After a safety call (2 weeks after baseline) they returned for identical assessments at week 8.
Groups:
- Memantine-1: Memantine: 10 mg bid
- Placebo-2: Matching placebo: bid
Period: Overall Study
Arm/Group | Memantine-1 | Placebo-2
Started | 20 | 20
Completed | 16 | 20
Not Completed | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Parallel Assignment Design. Patients were randomized for treatment with memantine or placebo, titrated over 4 weeks. UPDRS section I or II (primary endpoint), then Epworth sleepiness scale, fatigue severity scale, Hamilton depression scale, or Conner adult inventory secondary endpoints at end of treatment periods for both drug and placebo.
Groups:
- Memantine-1: Memantine: 10mg bid
- Total: Total of all reporting groups
Arm/Group | Memantine-1 | Placebo-2 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 14 | 14 | 28
Sex: Female, Male [Count of Participants; unit: Participants] — 16 female/24 male all groups
  Participants
    Female | 8 | 8 | 16
    Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson Disease Rating Scale (UPDRS).
Description: Assess the overall change from baseline in ON state motor United Parkinson Disease Rating scale (UPDRS) scores as assessed in the scale. The minimum score is 0 and the maximum score 199. The maximum score of 199 means the worst possible disability from Parkinson's Disease.
Time Frame: Baseline and 16 weeks
Population: Tabulations and univariate statistics on difference scores between visits were run using Intercooled Stata V8.0 and included Student's t-test with equal variances and contingency table analysis using Pearson's Chi-square test. Statistics were done using LOCF.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Memantine-1 | Placebo-2
Number analyzed (Participants) | 20 | 20
units on a scale
  Before treatment | 12 [6 to 30] | 12 [6 to 35]
  After treatment | 10 [7 to 28] | 10 [7 to 33]

2. Secondary Outcome: Analyses Will be Computed for the Categorical Dependent Variable (DV): Global Tremor Assessment by Examiner
Description: Change from baseline to end of study in the following assessment: global tremor assessment by examiner. The maximum total score is 48 and would indicate a high prevalence of tremor. The minimum total score is 0 and would indicate no tremor.
Time Frame: Baseline and 16 weeks
Population: Tabulations and univariate statistics on difference scores between visits were run using Intercooled Stata V8.0 for windows (Stata Corporation, College Station, Texas 77845), and included Student's t-test with equal variances and contingency table analysis using Pearson's Chi-square test. Statistics were done using LOCF. Corrections for multiple comparisons were not done.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Memantine-1 | Placebo-2
Number analyzed (Participants) | 20 | 20
scores on a scale
  Baseline | 2.8 (0.54) | 2.8 (0.54)
  16 Weeks | 2.8 (0.54) | 2.8 (0.54)

ADVERSE EVENTS:
Time Frame: Consent to end of study (24 weeks)
Description: The number of participants at risk for All-Cause Morality is 40, though most Parkinson's Disease patient do not die from Parkinson's Disease, they die from additional symptoms that develop.
Groups:
- Experimental: 1-Active Study Drug Memantine 10 mg Big: Memantine: 10 mg bid
- Placebo Comparator: 2-placebo Comparator: Matching placebo: bid
Arm/Group | Experimental: 1-Active Study Drug Memantine 10 mg Big | Placebo Comparator: 2-placebo Comparator
All-Cause Mortality (participants affected / at risk) | 3/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: 1-Active Study Drug Memantine 10 mg Big (N=20) | Placebo Comparator: 2-placebo Comparator (N=20)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
lethargy (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less